CLINICAL TRIAL: NCT06305637
Title: A Multi-center, Double-blind, Randomized, Placebo Controlled, Parallel-group Study, Comparing Ketoconazole Shampoo, 2% to Ketoconazole Shampoo, 2% (RS) and Both Active Treatments to a Placebo Control in the Treatment of Tinea Versicolor.
Brief Title: A Study Comparing Ketoconazole Shampoo, 2% and Ketoconazole 2% Shampoo (RS) in the Treatment of Tinea Versicolor.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sun Pharmaceutical Industries, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KTCS-2302
Record Dates: First submitted 2024-03-05; First posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Tinea Versicolor
MeSH Terms: conditions — Tinea Versicolor | interventions — Reference Standards

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Ketoconazole Shampoo, 2% (Experimental): The investigational product was applied on a single occasion topically to the damp skin of the affected area and a wide margin surrounding this area for 5 minutes and then rinsed off with water.
  Interventions: Drug: Ketoconazole Shampoo, 2%
- Ketoconazole Shampoo, 2% (Reference Standard) (Active Comparator): The investigational product was applied on a single occasion topically to the damp skin of the affected area and a wide margin surrounding this area for 5 minutes and then rinsed off with water.
  Interventions: Drug: Ketoconazole Shampoo, 2% (Reference Standard)
- Placebo Control (Placebo Comparator): The investigational product was applied on a single occasion topically to the damp skin of the affected area and a wide margin surrounding this area for 5 minutes and then rinsed off with water.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ketoconazole Shampoo, 2% — The investigational product was applied on a single occasion topically to the damp skin of the affected area and a wide margin surrounding this area for 5 minutes and then rinsed off with water.
  Other Names: Test Product
  Arms: Ketoconazole Shampoo, 2%
Drug: Ketoconazole Shampoo, 2% (Reference Standard) — The investigational product was applied on a single occasion topically to the damp skin of the affected area and a wide margin surrounding this area for 5 minutes and then rinsed off with water.
  Other Names: Reference Product
  Arms: Ketoconazole Shampoo, 2% (Reference Standard)
Drug: Placebo — The investigational product was applied on a single occasion topically to the damp skin of the affected area and a wide margin surrounding this area for 5 minutes and then rinsed off with water.
  Other Names: Vehicle
  Arms: Placebo Control

SUMMARY:
To demonstrate the efficacy, therapeutic equivalence and safety of Ketoconazole Shampoo, 2% (Taro Pharmaceuticals U.S.A., Inc.) and Ketoconazole 2% Shampoo (Reference Standard) in the treatment of tinea versicolor.

DETAILED DESCRIPTION:
A multi-center, double-blind, randomized, placebo controlled, parallel-group study, comparing Ketoconazole Shampoo, 2% (Taro Pharmaceuticals U.S.A, Inc.) to Ketoconazole Shampoo, 2% (Reference Standard) and both active treatments to a placebo control in the treatment of tinea versicolor.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or non-pregnant female aged ≥ 18 years
2. Subjects must have provided IRB approved written informed consent.
3. Subjects must have clinical diagnosis of tinea versicolor.
4. Subjects must be willing to refrain from using all other tinea versicolor medications or antifungals during the study, other than the investigational product.
5. Female Subjects of childbearing potential (excluding women who are premenarchal, surgically sterilized (by hysterectomy) or postmenopausal for at least 1 year), in addition to having a negative urine pregnancy test, must be willing to use an acceptable form of birth control during the study from the day of the first dose administration to 30 days after the last administration of study drug.

Exclusion Criteria:

1. Female Subjects who are pregnant, nursing or planning to become pregnant during study participation.
2. Subjects with a history of hypersensitivity or allergy to ketoconazole, other imidazole antifungals, and/or any of the study medication ingredients.
3. Subjects with the presence of any skin condition that would interfere with the diagnosis or assessment of tinea versicolor (e.g., vitiligo, pityriasis alba, post inflammatory hypopigmentation and hyperpigmentation, seborrheic dermatitis, pityriasis rosea, guttate psoriasis, tinea corporis, nummular eczema, secondary syphilis, confluent reticulated papillomatosis of Gougerot and Carteaud, and mycosis fungoides).
4. Treatment for tinea versicolor within the past 6 months that had been unresponsive to prescription topical or oral antifungals.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 430 (Actual)
Dates: Start 2023-12-04 (Actual); Primary Completion 2024-02-10 (Actual); Study Completion 2024-02-10 (Actual)

PRIMARY OUTCOMES:
To demonstrate the therapeutic equivalence and safety of the Investigational Product | Day 28 Visit
  Proportion of subjects with treatment success/cure

CONTACTS AND LOCATIONS:
Overall Officials: Natalie Yantovskiy, Study Director — Taro Pharmaceuticals, Inc.
Locations (1):
- Taro, Hawthorne, New York, United States

IPD SHARING:
Plan to Share IPD: No